CLINICAL TRIAL: NCT05956964
Title: Effects of Unloading and Sleep Restriction on Balance Regulation and Quadriceps Structure and Contractile Function
Brief Title: NM Balance Regulation With ULLS and Loss of Sleep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lance Bollinger (Other)
Collaborators: National Aeronautics and Space Administration (NASA) (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Lance Bollinger, Associate Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 84290; 80NSSC20M004 (Other Grant/Funding Number: NASA Kentucky)
Record Dates: First submitted 2023-07-03; First posted 2023-07-24 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Muscle Weakness; Quadriceps Muscle Atrophy; Sleep Disturbance
Keywords: sleep restriction; spaceflight; unweighting; posture
MeSH Terms: conditions — Muscle Weakness; Parasomnias

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to different arms via a matched-pairs design using the following criteria: age, sex, and race. Within each arm, the loaded limb will serve as an internal control to assess effects of unloading.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep Restriction (SR) (Experimental): The research team will provide participants with a pair of shoes to wear throughout the study. The right shoe will be modified to include a 5cm (approximately 2") rocker-style platform which will keep the left leg suspended during walking. Participants will also be provided with a pair of short crutches to assist with walking. Participants in the SR group will sleep only 5 hours for three consecutive nights.
  Interventions: Behavioral: Sleep Restriction
- Sleep Adequate (SA) (Active Comparator): The research team will provide participants with a pair of shoes to wear throughout the study. The right shoe will be modified to include a 5cm (approximately 2") rocker-style platform which will keep the left leg suspended during walking. Participants will also be provided with a pair of short crutches to assist with walking. Participants in the SA group will sleep for 9 hours for three consecutive nights.
  Interventions: Behavioral: Sleep Adequate

INTERVENTIONS:
Behavioral: Sleep Restriction — 5 hours of sleep for 3 days
  Arms: Sleep Restriction (SR)
Behavioral: Sleep Adequate — 9 hours of sleep for 3 days
  Arms: Sleep Adequate (SA)

SUMMARY:
The goal of this trial is to learn about how restricted sleep and not bearing weight on the leg affects muscle strength and posture control. Participants will walk exclusively on one leg, sleep at differing intervals, and complete posture tests, muscle strength tests, and muscle imaging. Researchers will compare adequate sleep and restricted sleep to see if muscle strength and posture are affected.

DETAILED DESCRIPTION:
During space flight, astronauts experience multiple physiological stimuli (such as microgravity and altered sleep cycles) which independently impair balance and strength. The goal of this project is to determine how these stimuli interact to affect static single-leg balance, balance during dynamic tasks, and muscle recruitment, strength, and remodeling.

Subjects (healthy adults age 18-50) will complete 13 days of unilateral lower limb suspension (ULLS, the gold standard analog for measuring space flight in ambulatory subjects). For the final three days of the study, subjects will be randomly assigned (via a matched pairs approach) to either normal sleep (7-9 hours per night) or restricted sleep (5 hours per night). Before and after the study, subjects will complete balance assessments and measures of muscle strength and recruitment. At the end of the study, subjects will also undergo diffusion tensor imaging for the thighs.

Balance testing will be conducted by examining sway in center of gravity during single leg stance and when stepping down from a box. Muscle strength and recruitment will be assessed via submaximal and maximal voluntary isometric contractions. Additionally, an interpolated twitch experiment will be performed to assess muscle recruitment and twitch properties. Diffusion Tensor imaging will be used to quantify muscle size and structure.

As prophylactic treatment against deep vein thrombosis (the major risk of ULLS), subjects will take an aspirin (81mg daily), wear compression stockings, complete passive range of motion exercises, and use intermittent pneumatic compression devices during sedentary times.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 50 years
* Regularly engaging in aerobic exercise (> 150min/wk) and resistance exercise (>1 time per week) for the past 12 months
* Regularly sleep at least 7 hours per night

Exclusion Criteria:

* Age < 18 or > 50 years
* Height between <150 (F) or <170 (M) and > 190 cm (both sexes)
* Waist circumference < 55cm or > 90cm (F) and < 75cm or > 100cm (M)
* Body mass index < 18.5 or > 27.5
* Do not regularly sleep between 7 and 9 hours each night
* Have a known sleep disorder
* Not regularly engaging in exercise for previous 12 months
* Blood clotting disorder
* Heart arrhythmia
* Implanted device which could negatively be affected by electrical impulse or strong magnetic field such as pacemaker, internal defibrillator, or cochlear implant
* Diagnosed cardiovascular, pulmonary, renal, or metabolic disease
* Pregnancy (within previous 6 months)
* Oral contraceptive use (within previous three months)
* High resting blood pressure (>140 systolic and/or > 90 diastolic)
* Currently or previously undergone gender-affirming therapy (hormone therapy or sexual reassignment surgery)
* Low back or leg injury in previous 6 months
* Currently taking medication to assist with sleep
* Muscle, bone, or joint injury that limits physical activity within previous 6 months
* Neurological disorder which affects balance (such as multiple sclerosis or Parkinson's disease)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2023-08-10 (Actual); Primary Completion 2025-03-14 (Actual); Study Completion 2025-03-14 (Actual)

PRIMARY OUTCOMES:
Change in Interpolated Twitch | Baseline and study completion, approximately 14 days
  Subjects will sit upright in an isokinetic dynamometer with the knee at 60° flexion. Gel electrode pads will be placed over the femoral nerve and just proximal to the patellar tendon. Square wave, constant current, doublet pulses from an electrical stimulator will be used to evoke twitches prior to, during, and following a maximal voluntary isometric contraction (MVIC).
Change in Single Leg Stand (SLS) | Baseline and study completion, approximately 14 days
  Balance will be assessed using a dual force plate system. Participants will be asked to stand on one leg and maintain their balance for 15 seconds
Muscle volume | Post-intervention, approximately 14 days after start of study
  Diffusion Tensor Imaging (DTI) will be used to quantify muscle volume. Subjects will lay supine, and slightly flex the knee (~10°) to elongate and straighten the quadriceps. A spine array coil will be placed on the MR-scanner table and a flexible body coil wrapped around the upper thigh and centered over mid-thigh of the dominant leg. Multiple images will be taken. DSI Studio program will be used to analyze raw images.
Change in Single Leg Land and Hold | Baseline and study completion, approximately 14 days
  Balance will be assessed using a dual force plate system. Participants will step off a wooden platform and land with one leg only in the middle of the respective force plate. As soon as the participant lands, they will be asked to maintain their position for 10 seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Lance Bollinger, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

DOCUMENTS (1):
  • Informed Consent Form (2024-04-24): https://cdn.clinicaltrials.gov/large-docs/64/NCT05956964/ICF_000.pdf